CLINICAL TRIAL: NCT04941872
Title: Comparison of 68Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2 PET/CT in Patients With Various Types of Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XMYY-2020KY042
Record Dates: First submitted 2021-06-20; First posted 2021-06-28 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2021-06

CONDITIONS: Tumor, Solid, FAPI, PET/CT, Metastasis
Keywords: Diagnosis, Tumor, Solid, FAPI, PET/CT, Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Disease

STUDY DESIGN:
Intervention Model Description: Subjects with various types of cancer undergo contemporaneous 68Ga-DOTA-2P(FAPI)2 and 68Ga-DOTA-FAPI-46 PET/CT either for an initial assessment or for recurrence detection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTA-2P(FAPI)2 PET/CT (Experimental): Each subject receive a single intravenous injection of and 68Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2, and undergo PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: 68Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2 PET/CT — Each subject receive a single intravenous injection of 68Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2, and undergo PET/CT imaging within the specified time.

SUMMARY:
To evaluate the potential usefulness of 68Ga-DOTA-2P(FAPI)2 positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various types of cancer, compared with 68Ga-DOTA-FAPI-46 PET/CT.

DETAILED DESCRIPTION:
In order to enhance the tumor uptake and tumor retention time, we designed the dimer structure of fibroblast activation protein inhibitor (FAPI), a novel imaging agent that targeting cancer-associated fibroblasts expressed in various types of cancer, 68Ga-DOTA-2P(FAPI)2. Subjects with various types of cancer underwent contemporaneous 68Ga-DOTA-2P(FAPI)2 and 68Ga-DOTA-FAPI-46 PET/CT either for an initial assessment or for recurrence detection. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 68Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2 PET/CT were calculated and compared to evaluate the diagnostic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* (i) adult patients (aged 18 years or order);
* (ii) patients with suspected or newly diagnosed or previously treated malignant tumors (supporting evidence may include magnetic resonance imaging (MRI), CT, tumor markers and pathology report);
* (iii) patients who had scheduled both 8Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2 PET/CT PET/CT scans;
* (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* (i) patients with non-malignant lesions;
* (ii) patients with pregnancy;
* (iii)the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of 68Ga-DOTA-FAPI-46 / 68Ga-DOTA-2P(FAPI)2 for each primary tumor of subject or suspected lymph metastasis.

SECONDARY OUTCOMES:
Sensitivity | 30 days
  The sensitivity of 68Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2 PET/CT
Specificity | 30 days
  The specificity of 68Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2 PET/CT
The positive predictive value (PPV) | 30 days
  The positive predictive value (PPV) of 68Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2 PET/CT
The negative predictive value (NPV) | 30 days
  The negative predictive value (NPV) of 68Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2 PET/CT
The accuracy | 30 days
  The accuracy of 68Ga-DOTA-FAPI-46 and 68Ga-DOTA-2P(FAPI)2 PET/CT
Radiation Dosimetry | 30 days
  Mean absorbed radiation doses were estimated using the source and target organ framework. Five patients with different cancers underwent serial 68Ga-DOTA-2P(FAPI)2 PET/CT scans at three time points following radiotracer injection: 10 minutes, 1 hour, and 3 hours. The source organs consisted of the kidneys, bladder, liver, heart, spleen, bone marrow, uterus, and body remainder. OLINDA/EXM software was used to fit and integrate the kinetic organ activity data to yield total body and organ time-integrated activity coefficients/residence times and finally organ absorbed doses.

CONTACTS AND LOCATIONS:
Overall Officials: Long Sun, PhD, Study Director — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First affiliated hospital of xiamen university, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No